CLINICAL TRIAL: NCT00003610
Title: Phase III Comparison of Oral Capsaicin Lozenge Versus Placebo Lozenge for Radiation-Induced Mucositis
Brief Title: Capsaicin Lozenges in Treating Patients With Mucositis Caused by Radiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-969257; CDR0000066687 (Registry Identifier: PDQ (Physician Data Query)); NCI-P98-0136
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Head and Neck Cancer; Radiation Toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries | interventions — Capsaicin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- capsaicin + radiation therapy (Experimental): Patients receive one lozenge orally of capsaicin four times daily. Treatment begins within the first 3 days of radiation therapy and continues during and for two weeks after radiation therapy is completed.
  Interventions: Dietary Supplement: capsaicin; Radiation: radiation therapy
- placebo + radiation therapy (Placebo Comparator): Patients receive one lozenge orally of placebo four times daily. Treatment begins within the first 3 days of radiation therapy and continues during and for two weeks after radiation therapy is completed.
  Interventions: Other: placebo; Radiation: radiation therapy

INTERVENTIONS:
Dietary Supplement: capsaicin
  Arms: capsaicin + radiation therapy
Other: placebo
  Arms: placebo + radiation therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Capsaicin lozenges may be effective treatment for mucositis caused by radiation therapy. It is not yet known whether capsaicin lozenges are more effective than no treatment for mucositis caused by radiation therapy.

PURPOSE: Randomized phase III trial to study the effectiveness of capsaicin lozenges in treating patients with mucositis caused by radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of capsaicin lozenges in terms of frequency, duration, and severity of mouth pain caused by radiation therapy to the oral cavity. II. Evaluate the toxicity of this regimen in these patients.

OUTLINE: This is a randomized, double blind, placebo controlled study. Patients are stratified according to dentures (yes vs no), smoking history (none vs currently vs past only), radiation therapy (primary vs postoperative adjuvant), planned radiation dose (5000-6000 cGy vs greater than 6000 cGy), planned fluoride use (yes vs no), and amount of oral mucosa in radiation field (one- to two-thirds vs greater than two-thirds). Patients receive one lozenge orally of capsaicin or placebo four times daily. Treatment begins within the first 3 days of radiation therapy and continues during and for two weeks after radiation therapy is completed.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Scheduled to receive radiation treatment to at least one third of the oral cavity at a total dose of at least 5000 cGy using 200 cGy/fraction Must be entered on study within first 3 days of radiation No open mouth sores at study entry

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No known intolerance to capsaicin No allergy to citric acid, cherry flavorings, or FC and C red dye #3 or #40

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the oral mucosa Surgery: Not specified Other: No requirement for tube feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1998-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
frequency of mouth pain | Up to 2 weeks post-radiation treatment
duration of mouth pain | Up to 2 weeks post-radiation treatment
severity of mouth pain | Up to 2 weeks post-radiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Scott Okuno, MD, Study Chair — Mayo Clinic
Locations (17):
- United States (17):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota